CLINICAL TRIAL: NCT02812433
Title: Sildenafil Administration to Treat Neonatal Encephalopathy (SANE) and Repair Brain Injury Secondary to Birth Asphyxia: A Randomized, Double-blind, Placebo-controlled Pilot Phase Ib Study
Brief Title: Sildenafil Administration to Treat Neonatal Encephalopathy
Acronym: SANE-01
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Pia Wintermark, Assistant Professor of Paediatrics, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SANE-01
Record Dates: First submitted 2016-06-19; First posted 2016-06-24 (Estimated); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Neonatal Encephalopathy
Keywords: birth asphyxia; brain; hypoxic-ischemic encephalopathy; neonate; neuroprotection; neurorestoration; newborn; sildenafil
MeSH Terms: conditions — Asphyxia Neonatorum; Hypoxia-Ischemia, Brain | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sildenafil (Active Comparator): Sildenafil 2 mg/kg/dose per os twice a day for seven consecutive days (from day 2 of life to day 9 of life) if brain injury on day 2 of life
  Interventions: Drug: Sildenafil
- Ora-Blend (Placebo Comparator): Ora-Blend 2 mg/kg/dose per os twice a day for seven consecutive days (from day 2 of life to day 9 of life) if brain injury on day 2 of life
  Interventions: Drug: Ora-Blend

INTERVENTIONS:
Drug: Sildenafil — sildenafil 2 mg/kg/dose per os twice a day for seven consecutive days (from day 2 of life to day 9 of life) if brain injury on day 2 of life
  Arms: Sildenafil
Drug: Ora-Blend — Ora-Blend, 2 mg/kg/dose per os twice a day for seven consecutive days (from day 2 of life to day 9 of life) if brain injury on day 2 of life
  Arms: Ora-Blend

SUMMARY:
Despite improvements in neonatal care, birth asphyxia in term newborns remains a serious condition causing significant mortality and long-term morbidity, including cerebral palsy and mental retardation. Currently, no treatment exists to repair brain injuries secondary to neonatal asphyxia. The only available treatment for this condition is hypothermia that may prevent but not repair the development of brain injury. The success of this therapy is limited.

Sildenafil already is used with some newborns for other purposes (i.e., persistent pulmonary hypertension), but, surprisingly, its effect on the newborn brain has never been studied systematically. The findings of the investigators in the rat model of term neonatal encephalopathy demonstrated that the administration of sildenafil following asphyxia promotes brain injury recovery. Thus, the investigators hypothesize that sildenafil may improve neurodevelopmental outcome in term asphyxiated newborns, in whom hypothermia treatment has failed to prevent the development of brain injury.

DETAILED DESCRIPTION:
Before being able to run a large multicenter randomized trial to prove this hypothesis, the investigators need to run a phase Ib pilot trial to ensure the feasibility and safety of using sildenafil in this population of newborns. Thus, for this phase Ib study, the investigators hypothesize that sildenafil can be safely used with term asphyxiated newborns treated with hypothermia. The investigators will test this hypothesis with the following specific aims:

1. Safety (primary): ensure that sildenafil can be safely used in asphyxiated newborns treated with hypothermia;
2. Tolerability (secondary): study the pharmacokinetics and pharmacodynamics of sildenafil in these newborns;
3. Efficacy (exploratory): determine whether sildenafil improves neurodevelopment at 2 years of age, decreases brain injury on day 30 of life and decreases neuroinflammation.

ELIGIBILITY:
Inclusion Criteria:

* Male and female asphyxiated newborns meeting the criteria for induced hypothermia:

  * Gestational age ≥ 36 weeks and birth weight ≥ 1800 g
  * Evidence of fetal distress, such as a history of an acute perinatal event, a cord pH ≤ 7.0 or base deficit ≤ - 16 mEq/L
  * Evidence of neonatal distress, such as an Apgar score ≤ 5 at 10 minutes, a postnatal blood gas pH obtained within the first hour of life ≤ 7.0 or base deficit ≤ - 16 mEq/L, or a continued need for ventilation initiated at birth and continued for at least 10 minutes
  * Evidence of moderate to severe neonatal encephalopathy by an abnormal neurological exam and/or an amplitude-integrated electroencephalogram (aEEG) These newborns will receive whole-body cooling to an esophageal temperature of 33.5°C, initiated within the first 6 hours of life, continued for 72 hours, and then they were slowly rewarmed using standard protocol .
* Evidence on a brain MRI performed on day 2 of life (while they are treated with hypothermia) of any type of brain parenchymal injury patterns typically encountered in asphyxiated newborns.

If they meet the criteria for hypothermia treatment and demonstrate brain injury on day 2 of life, they will be randomized to sildenafil or placebo treatment.

Exclusion Criteria:

* Newborns with complex congenital heart disease
* Newborns with cerebral malformations
* Newborns with genetic syndrome
* Newborns with intraventricular and/or intraparenchymal hemorrhage on the MRI performed on day 2 of life
* Moribund infants not expected to survive

Ages: 0 Minutes to 48 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2022-01 (Actual)

PRIMARY OUTCOMES:
Serious adverse events | Day 1 to 14 of life
  Close monitoring for adverse events such as death, hypotension, persistent pulmonary hypertension, altered renal or hepatic function, etc to assess the safety of sildenafil

SECONDARY OUTCOMES:
Plasmatic concentrations of sildenafil and N-desmethyl sildenafil | Day 2 to 10 of life
  To determine the tolerability of sildenafil (pharmacokinetics/pharmacodynamics)

OTHER OUTCOMES:
Brain injury severity as per a previously described brain injury score | Day 30 of life, compared to day 2 of life
  Exploratory outcome to explore efficacy (brain injury)
panel of 45 inflammatory biomarkers known to be involved in neuroinflammation, including interleukin-1 (IL-1) alpha and its receptor, interleukin-6 (IL-6) and tumor necrosis factor (TNF) alpha | Day 2 to 30 of life
  Exploratory outcome to explore efficacy (neuroinflammation)
Bayley Scale of Infant Development (BSID-III) | 1 year and 2 years of age
  Exploratory outcome to explore efficacy (neurodevelopment)

CONTACTS AND LOCATIONS:
Overall Officials: Pia Wintermark, Pia, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- Montreal Children's Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wintermark P, Lapointe A, Steinhorn R, Rampakakis E, Burhenne J, Meid AD, Bajraktari-Sylejmani G, Khairy M, Altit G, Adamo MT, Poccia A, Gilbert G, Saint-Martin C, Toffoli D, Vachon J, Hailu E, Colin P, Haefeli WE. Feasibility and Safety of Sildenafil to Repair Brain Injury Secondary to Birth Asphyxia (SANE-01): A Randomized, Double-blind, Placebo-controlled Phase Ib Clinical Trial. J Pediatr. 2024 Mar;266:113879. doi: 10.1016/j.jpeds.2023.113879. Epub 2023 Dec 22. PMID 38142044
- See also: Related Info — http://www.neobrainlab.org